CLINICAL TRIAL: NCT01773746
Title: The Premature Infants Resuscitated With Oxygen or Air (PRESOX) Trial
Brief Title: Study of Room Air Versus 60% Oxygen for Resuscitation of Premature Infants
Acronym: PRESOX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor Recruitment
Sponsor: Sharp HealthCare (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Neil Finer, Clinical Consultant, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-3602
Record Dates: First submitted 2013-01-10; First posted 2013-01-23 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Extreme Prematurity - Less Than 28 Weeks
Keywords: neonatal; resuscitation; room air

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Room Air (Active Comparator): Neonatal Resuscitation using continuous positive airway pressure(CPAP) or positive pressure ventilation (PPV) will be provided with 21% oxygen. Infants will remain on 21% oxygen until they have a functioning oximeter when SpO2 will be managed as below. FiO2 will be increased by 10% increments when the infant's SpO2 is below the lower sat limit for 30 seconds and repeated if the SpO2 remains outside the limit for a subsequent interval of 30 seconds as often as is necessary to bring the SpO2 within the pre-specified range. The FiO2 will be decreased by 10% increments when the SpO2 is above the upper limit for 30 seconds and repeated if the SpO2 remains outside the limit for a subsequent interval of 30 second as often as is necessary to bring the SpO2 within the pre-specified range.
  Interventions: Other: Neonatal Resuscitation
- 60% Group (Active Comparator): Neonatal Resuscitation using CPAP or PPV will be provided with 60% oxygen. Infants will remain on 60% oxygen until they have a functioning oximeter at which time their SpO2 will be managed as described below FiO2 will be increased by 10% increments when the infant's SpO2 is below the lower sat limit for 30 seconds and repeated if the SpO2 remains outside the limit for a subsequent interval of 30 seconds as often as is necessary to bring the SpO2 within the pre-specified range. The FiO2 will be decreased by 10% increments when the SpO2 is above the upper limit for 30 seconds and repeated if the SpO2 remains outside the limit for a subsequent interval of 30 second as often as is necessary to bring the SpO2 within the pre-specified range.
  Interventions: Other: Neonatal Resuscitation

INTERVENTIONS:
Other: Neonatal Resuscitation — CPAP or Positive Pressure Ventilation will be provided.

SUMMARY:
The most appropriate initial oxygen concentration for the resuscitation of the extremely low birth weight infant has not been established using large well designed, randomized, blinded, prospective trials and the level of oxygen utilized by practitioners in this situation is highly variable. This proposed trial will use targeted oxygen saturation levels over the first 15 to 20 minutes of life to compare a low and a higher initial oxygen level for the resuscitation of such infants, and will be large enough to evaluate short term outcomes of survival without oxygen at 36 weeks and survival without retinopathy of prematurity, and the long term outcome of survival without significant neurodevelopmental impairment at 2 years of age. Such information is urgently required to provide an evidence basis for the initial oxygen concentration for resuscitation of these very preterm infants.

DETAILED DESCRIPTION:
The Premature Infants Resuscitated with Oxygen or Air (PRESOX) trial, is a prospective randomized clinical trial of extremely premature infants that will assess the use of a low and high oxygen concentration for the initial resuscitation. The hypothesis is that infants resuscitated with a lower oxygen concentration at birth will have a increase in survival without bronchopulmonary dysplasia (BPD) or retinopathy of prematurity (ROP) during their initial hospitalization, and will have a increase in survival without neurodevelopmental impairments.

Previous studies of mostly term newborn infants have demonstrated that initial resuscitation with room air compared to 100% oxygen resulted in improved outcomes and an overall decrease in mortality. The analysis of these studies demonstrated that the reduction in mortality was very significant in the preterm infants that had been included in these trials. A number of small clinical trials have now demonstrated that it is feasible to treat very preterm infants with lower versus higher concentrations of oxygen while carefully monitoring their oxygen saturation in the minutes following delivery. As review of the previous observations demonstrated that there was a reduction in death using lower oxygen concentration, it is imperative that a large study of preterm infants be conducted to determine if a lower compared to a higher oxygen concentration for the initial resuscitation will lead to improved short and longer term outcomes including survival without neurodevelopmental disability.

The PRESOX trial will randomize infants from 23 weeks gestation to 28 weeks gestation who require resuscitation at birth to receive either room air or 60% oxygen. Oxygen saturation will be monitored from the first minute of life and the initial oxygen concentration will be titrated using a unique purpose built device which will track the oxygen saturation (SpO2) within the chosen target limits. The targets chosen allow the infants oxygen saturation to follow the increase seen in normal preterm infants who do not require resuscitation. Following resuscitation the infants will be transferred to the Neonatal Intensive Care Unit and management will follow the usual care in those units. In a subset of infants, levels of antioxidants from the infant's blood and urine will be measured by Dr M Vento. This portion of the study is already funded by the combined Spanish Ministries of Health and Science. Antioxidants are known to increase with exposure to oxygen. The infants will return for a neurodevelopmental follow up examination at the age of two years.

This trial will provide urgently needed evidence to establish the most optimal care to these very fragile preterm infants.

ELIGIBILITY:
Inclusion Criteria:

Infants with a gestational age of 23 0/7 to 28 6/7 weeks by best obstetrical estimate.

Infants who will receive full resuscitation as necessary, i.e., no parental request or physician decision to forego resuscitation Infants whose parents/legal guardians have provided consent for enrollment, or for whom a waiver of consent is in place Infants without known major congenital malformations prior to delivery

Exclusion Criteria:

Any infant transported to the center after delivery Infants whose parents/legal guardians refuse consent Infants born when the research apparatus/study personnel are not available Infants < 23 weeks 0 days or > 28 weeks 6 days, completed weeks of gestation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-08; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Survival with neurodevelopmental impairment | 18-22 mos.
  To determine if resuscitation starting with 21% oxygen and a targeted SpO2 strategy will increase survival without significant neurodevelopmental impairment at 18 to 22 months when compared with starting with 60% oxygen and a targeted SpO2 strategy.

SECONDARY OUTCOMES:
Survival without bronchopulmonary dysplasia | 36 weeks
  2. To determine if resuscitation of extremely low gestational age neonates (ELGAN) starting with 21% oxygen and a targeted SpO2 strategy will increase survival without bronchopulmonary dysplasia when compared with starting with 60% oxygen and a targeted SpO2 strategy.
Survival without ROP | 36 weeks
  3. To determine if resuscitation of extremely low gestational age neonates (ELGAN) starting with 21% oxygen and a targeted SpO2 strategy will increase survival without Retinopathy of Prematurity when compared with starting with 60% oxygen and a targeted SpO2 strategy.
Decreased GSSG/GSH Ratio | Birth,1,3,7 days
  4. To determine if resuscitation starting with 21% oxygen and a targeted SpO2 strategy will result in decreased GSSG/GSH ratio concentrations and decreased production of isofurans when compared with starting with 60% oxygen and a targeted SpO2 strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Neil N Finer, MD, Principal Investigator — UCSD Medical Center; Maximo Vento, MD, Principal Investigator — Hospital La Fe, Valencia Spain; Ola D Saugstad, MD, PhD, Principal Investigator — The National Hospital, Oslo Norway
Locations (22):
- United States (6):
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California
  - Connecticut Children's Medical Center, Farmington, Connecticut
  - University of Miami Miller School of Medicine, Miami, Florida
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - OU - Tulsa - Saint Francis Hospital, Tulsa, Oklahoma
- Austria (2):
  - Innsbruck Medical University, Innsbruck
  - Medical University of Vienna, Vienna
- Chu-Toulouse, Toulouse, France
- Ulm University, Ulm, Germany
- National Maternity Hospital, Dublin, Ireland
- Italy (2):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - University of Siena, Siena
- Poznan University of Medical Sciences, Poznan, Poland
- St. Petersberg State Pediatric Medical University, Saint Petersberg, Russia
- University Medical Center Ljubljana, Ljubljana, Slovenia
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Saint Joan de Deu, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital La Fe, Valencia
- Karolinska Institutet, Stockholm, Sweden
- James Cook University Hospital, Middlesbrough, United Kingdom